CLINICAL TRIAL: NCT05856825
Title: Long-Term Outcomes of Robot-Assisted Radical Cystectomy: A Real-World Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2021-322
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Bladder Cancer; Robot-assisted Radical Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (32):
- Sun Yat-sen Memorial Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy
- Renji Hospital, Shanghai Jiaotong University School of Medicine
  Interventions: Procedure: Robot-assisted radical cystectomy
- The Third Medical Centre of Chinese PLA General Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy
- The First Affiliated Hospital of Zhengzhou University
  Interventions: Procedure: Robot-assisted radical cystectomy
- Zhejiang Provincial People's Hospital, Affiliated People's Hospital, Hangzhou Medical College
  Interventions: Procedure: Robot-assisted radical cystectomy
- Southwest Hospital, Third Military Medical Hospital (Army Medical University)
  Interventions: Procedure: Robot-assisted radical cystectomy
- Tongji Hospital Affiliated to Tongji Medical College Hust
  Interventions: Procedure: Robot-assisted radical cystectomy
- The First Affiliated Hospital of Xi'an Jiaotong University
  Interventions: Procedure: Robot-assisted radical cystectomy
- The First Affiliated Hospital of Navy Medical University
  Interventions: Procedure: Robot-assisted radical cystectomy
- The First Affiliated Hospital of Nanchang University
  Interventions: Procedure: Robot-assisted radical cystectomy
- Zhongda Hospital Southeast University
  Interventions: Procedure: Robot-assisted radical cystectomy
- The Second Xiangya Hospital, Central South University
  Interventions: Procedure: Robot-assisted radical cystectomy
- The First Affiliated Hospital of Nanjing Medical University
  Interventions: Procedure: Robot-assisted radical cystectomy
- Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy
- Gansu Provincial Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy
- The Affiliated Yantai Yuhuangding Hospital of Qingdao University
  Interventions: Procedure: Robot-assisted radical cystectomy
- West China Hospital, Sichuan University
  Interventions: Procedure: Robot-assisted radical cystectomy
- The First Hospital of China Medical University
  Interventions: Procedure: Robot-assisted radical cystectomy
- The Third Xiangya Hospital of Central South University
  Interventions: Procedure: Robot-assisted radical cystectomy
- General Hospital of Central Theater Command
  Interventions: Procedure: Robot-assisted radical cystectomy
- Kunming First People's Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy
- The East Campus of Qingdao Municipal Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy
- The second Affiliated Hospital of Kunming Medical University
  Interventions: Procedure: Robot-assisted radical cystectomy
- Second Hospital of Dalian Medical University
  Interventions: Procedure: Robot-assisted radical cystectomy
- The Second Affiliated Hospital of Xi'an Jiaotong University
  Interventions: Procedure: Robot-assisted radical cystectomy
- The First Hospital of Jilin University
  Interventions: Procedure: Robot-assisted radical cystectomy
- Zhejiang Cancer Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy
- Peking University Third Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy
- Changzheng Hospital, Naval Medical University
  Interventions: Procedure: Robot-assisted radical cystectomy
- Peking Union Medical College Hospital
  Interventions: Procedure: Robot-assisted radical cystectomy
- The First Affiliated Hospital of Chongqing Medical University
  Interventions: Procedure: Robot-assisted radical cystectomy
- Beijing United Family Hospital and Clinics
  Interventions: Procedure: Robot-assisted radical cystectomy

INTERVENTIONS:
Procedure: Robot-assisted radical cystectomy — Robot-assisted radical cystectomy

SUMMARY:
A multicenter, retrospective research was conducted. Patients who underwent robot-assisted radical cystectomy (RARC) from for bladder cancer in 32 institutions in China were enrolled in this study. Baseline condition, perioperative, pathological, and survival outcome were collected. The study was aimed to report the real-world condition of RARC in China, and evaluate its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old; Clinical stage Ta-T4a/N0-3/M0.

Exclusion Criteria:

* Severe cardiovascular disease; history of previous major abdominopelvic surgery; patients with distant metastases; medical history of malignancy in other organs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent robot-assisted radical cystectomy for bladder cancer from 2012 to 2021 in 32 large medical institutions in China.
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Five years
  Time from surgery until death from any cause
Recurrence-free survival | Five years
  Time from surgery to tumor recurrence which identified either pathologically or radiographically
Cancer-specific survival | Five years
  Time from date of surgery to death due to bladder cancer

IPD SHARING:
Plan to Share IPD: No